CLINICAL TRIAL: NCT01879761
Title: Immune Resolution After Staphylococcus Aureus Bacteremia
Status: Active, not recruiting | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 13-0491
Record Dates: First submitted 2013-06-10; First posted 2013-06-18 (Estimated); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Immune Response To Sepsis; Staphylococcus Aureus Infection
Keywords: Immunosuppressed; Sepsis; Staphylococcus Aureus; Bacteremia; HLA-DR
MeSH Terms: conditions — Staphylococcal Infections; Sepsis; Bacteremia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Isolated monocytes from whole blood for HLA-DR measurement. Serum and plasma for cytokine measurements
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Immunosuppressed: Immunosuppressed includes patients with any one of the following:
  1. a diagnosis of a hematological malignancy
  2. a diagnosis of HIV
  3. myelosuppressive chemotherapy in the previous 90 days
  4. immune-modulating medications in the previous 90 days
- Non-Immunosuppressed: Subject does not fit immunosuppressed criteria

SUMMARY:
The purpose of this study is to determine how monocyte HLA-DR and other markers of immune function change with time in patients with and without prior immune dysfunction who survive sepsis from Staphylococcus aureus bacteremia.

We hypothesize that patients with prior immune dysfunction will have greater reductions in HLA-DR and other markers of immune function after an episode of sepsis than people who do not have prior immune dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* At least one blood culture positive for S. aureus
* Patients aged ≥18 years
* At least two of four systemic inflammatory response syndrome (SIRS) criteria on the day of positive blood cultures. SIRS criteria are:

  * Body temperature less than 36°C(96.8°F) or greater than 38°C(100.4°F)
  * Heart rate greater than 90 beats per minute
  * Tachypnea (high respiratory rate), with greater than 20 breaths per minute; or, an arterial partial pressure of carbon dioxide less than 32 mmHg
  * WBC less than 4000 cells/mm³ (4 x 109 cells/L) or greater than 12,000 cells/mm³ (12 x 109 cells/L); or the presence of greater than 10% immature neutrophils (band forms)

Exclusion Criteria:

* Sequential Organ Failure Assessment (SOFA) score > 12 on day of positive blood cultures
* Survival expected to be < 7 days from positive blood cultures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital inpatients with Staphylococcus aureus bacteremia who are over 18 years old.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2013-06; Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
HLA-DR and cytokines | 0-30 days
  Percent expression of HLA-DR on monocytes will be measured by flow cytometry. Cytokine levels will be measured by ELISA.

SECONDARY OUTCOMES:
New Infections | 0-90 days

OTHER OUTCOMES:
Mortality | 0-90 days

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chicago Hospital, Chicago, Illinois, United States